CLINICAL TRIAL: NCT05283980
Title: Pectoral Nerve Blocks (PECs) for Cardiovascular Implantable Electronic Device Placement: A Pilot Study
Brief Title: Pectoral Nerve Blocks (PECs) for Cardiovascular Implantable Electronic Device Placement
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Sankalp Sehgal, Instructor, Principal Investigator, Anesthesia Attending, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2021P001063
Record Dates: First submitted 2022-03-08; First posted 2022-03-17 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Pain, Postoperative; Pain, Acute; Pain, Chest; Pain; Satisfaction, Patient; Opioid Use, Unspecified; Opioids; Harmful Use
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Chest Pain; Pain; Patient Satisfaction | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: This is prospective, randomized, triple-blinded placebo-controlled study. Subjects will be randomize to undergo PECs block in the pre-procdure/ pre-operative area with either ).25% bupivacaine or 0.9% normal saline. They will then undergo the CIED placement in electrophysiology lab as current standard of care.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Enrolled subjects will be randomized to one of the two study groups, in a 1:1 randomization ratio. Patients randomized to Group 1, or the bupivacaine group, will receive up to 25cc of 0.25% bupivacaine hydrochloride for the PECs blocks. In Group 2, patients will receive up to 25cc of normal saline. Use of placebo is a standard control procedure in clinical trials and will allow for the assessment of unbiased quantitative data on the efficacy across all treatment groups.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bupivacaine Group (Experimental): Receive up to 25 ml of 0.25% bupivacaine hydrochloride for the Pecs block
  Interventions: Drug: 0.25% Bupivacaine
- Control group (Placebo Comparator): Receive up to 25 ml of normal 0.9% sodium chloride for the Pecs block
  Interventions: Drug: 0.25% Bupivacaine

INTERVENTIONS:
Drug: 0.25% Bupivacaine — The intervention group/ bupivacaine group will receive up to 25 ml of 0.25% bupivacaine hydrochloride for the Pecs block in comparison to the control group that would receive 0.9% normal saline

SUMMARY:
The purpose of this study is to determine whether administration of a pectoral nerve blocks (Pecs I and II) with 0.25% bupivacaine are more effective as compared to placebo to provide analgesia for cardiac implantable electronic device (CIED) placement in cardiac electrophysiology lab

DETAILED DESCRIPTION:
Cardiovascular implantable electrical device (CIED) is a generalized term for pacemakers, implantable cardiac devices (ICDs) and cardiac resynchronization therapy (CRT) devices. CRT is a modality of cardiac pacing that provides simultaneous pacing of left ventricle (LV) and right ventricle (RV) as biventricular (BiV) pacing (CRT-pacemaker or CRT-P), or by a combined CRT-implantable-defibrillator (CRT-D). The indication for pacemaker implantation in a patient is abnormal cardiac electrical conduction such as sinus node dysfunction or high-grade atrioventricular block. CRT is indicated for patients with symptomatic heart failure with left bundle branch block. Patients undergoing CIEDs often have multiple other associated comorbidities such as pulmonary disease, chronic kidney disease etc. which places them at a high-risk for undergoing these procedures.

Every year, more than 500,000 CIEDs are implanted in the United States alone. These procedures are being done with increasing frequency in patients with arrhythmias, heart failure and other risk factors for sudden cardiac death. Opioid prescription usage and persistent use of opioids after CIED procedures remains very high. In the context of current opioid crisis, there is a growing need to find alternatives to optimize pain and limit opioid usage in the patient population.

The current standard practice for CIED placement is either under monitored anesthesia care (MAC) or general anesthesia. MAC is sedation and is usually performed using benzodiazepines, opioids, and propofol. Deleterious effects of opioids during sedation include respiratory or hemodynamic compromise, particularly in this high-risk patient population with low reserve. General anesthesia is invasive requiring endotracheal intubation and positive pressure ventilation, which can also compromise cardiorespiratory function. Finally, some patients with obesity or obstructive sleep apnea may have low tolerance to sedation and opioid use in procedures involving tunneling of leads or deeper chest wall tissue dissection. Despite procedural sedation or general anesthesia, patients generally continue to require pain medications postoperatively due to residual pain from the procedure.

Nerve blocks involve injection of local anesthetic around peripheral nerves or their branches to interrupt pain and other sensory signals thus alleviating pain. Pectoralis or Pecs block is one such nerve block and has recently been effectively in increasing evidence for various surgeries and procedures on chest wall. Few case reports in adult population undergoing pacemaker, ICD and CRT placement also emphasize the utility of these blocks especially in patients who are critically ill. Preliminary studies have shown lower sedation requirements and higher patient and proceduralist satisfaction with use of PEC block in these patients.

Moreover, there is no large study has evaluated the utility of PECs block in this patient population undergoing CIED insertion and there remains a need to investigate their utility in a systematic study.

There are two components to a Pecs block: Pecs I block that targets the lateral and medial pectoral nerves, suppliying both pectoral muscles (major and minor, and Pecs II block that targets the anterior and lateral division of the thoracic intercostal nerves T2-T6, the long thoracic nerve (C5-C7) which supplies the serratus anterior muscle and the thoracodorsal nerve (C6-C8) which innervates the latissimus dorsi muscle. Thus, combination of both Pecs I and II blocks can provide a widespread analgesic coverage and has been previously studied for analgesia for breast surgeries and also in thoracic trauma. It is a promising option considering its efficacy and ease of administration and may prove to be a useful analgesic technique in patients undergoing CIED insertion or replacement. The block is devoid of the systemic adverse events associated with opioids and hemodynamic complications associated with general anesthesia. It is a relatively superficial block and is therefore safe even on patient on antiplatelet therapy. It could prove useful in reducing intra-procedure analgesic requirement in the acute setting of postoperative pain as well as preventing chronic pain and has the potential to become the standard of care for analgesia in CIED procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Undergoing CIED placement in electrophysiology lab
* Booked with anesthesia service for the procedure.

Exclusion Criteria:

* Current participation in another interventional study
* Use of mechanical circulatory support device
* Emergent procedures
* Patients receiving other modalities of regional anesthesia like intrathecal morphine
* Chronic opioid use for chronic pain conditions with tolerance (total daily dose of an opioid at or more than 30 mg morphine equivalent for more than one month within the past year)
* Current use of SSRI, TCA, anti-epileptics, gabapentin, or pregabalin as part of multimodal pain management
* Hypersensitivity to bupivacaine
* Hemodynamics related: Oxygenation outside of normal limits (defined as PaO2 < 60mmHg on an FiO2 of 1.0 or SpO2 < 85% within 30 minutes prior to drug administration), Received an infusion or bolus ≥ 0.05 mcg/kg/min of epinephrine o Received an infusion or bolus ≥ 0.50 mcg/kg/min of milrinone, Received an infusion or bolus ≥ 0.20 mcg/kg/min of norepinephrine o Significant clinician or nursing concern, Hemodynamically unstable (defined as HR > 120, SBP < 80, MAP < 50 within 30 minutes prior to drug administration)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | 24 hours peri-procedure
  peri-operative 24-hour consumption of opioids measured as OMEs (Opioid milliequivalents) in patients undergoing CIED procedures with and without Pecs blocks

SECONDARY OUTCOMES:
Pain scores on a scale 1 - 10, 1 being the least pain and 10 being the worst pain | at 1 hour, 12 hour and 24hours
  measure patient pain scores at 1 hour, 12 hours and 24hours after CIED procedure completion
Patient satisfaction scores | at 24 hours post-procedure
  compare patient satisfaction scores at 24 hours between the two study groups and report the incidence of overall complications

CONTACTS AND LOCATIONS:
Overall Officials: Sankalp Sehgal, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- BIDMC, Boston, Massachusetts, United States

REFERENCES:
- [Background] Yang JK, Char DS, Motonaga KS, Navaratnam M, Dubin AM, Trela A, Hanisch DG, McFadyen G, Chubb H, Goodyer WR, Ceresnak SR. Pectoral nerve blocks decrease postoperative pain and opioid use after pacemaker or implantable cardioverter-defibrillator placement in children. Heart Rhythm. 2020 Aug;17(8):1346-1353. doi: 10.1016/j.hrthm.2020.03.009. Epub 2020 Mar 20. PMID 32201270
- [Background] Fujiwara A, Komasawa N, Minami T. Pectoral nerves (PECS) and intercostal nerve block for cardiac resynchronization therapy device implantation. Springerplus. 2014 Aug 5;3:409. doi: 10.1186/2193-1801-3-409. eCollection 2014. PMID 25120950
- [Background] Mavarez AC, Ripat CI, Suarez MR. Pectoralis Plane Block for Pacemaker Insertion: A Successful Primary Anesthetic. Front Surg. 2019 Nov 20;6:64. doi: 10.3389/fsurg.2019.00064. eCollection 2019. PMID 31824958
- [Background] Froyshteter AB, Bhalla T, Tobias JD, Cambier GS, Mckee CT. Pectoralis blocks for insertion of an implantable cardioverter defibrillator in two patients with Duchenne muscular dystrophy. Saudi J Anaesth. 2018 Apr-Jun;12(2):324-327. doi: 10.4103/sja.SJA_624_17. PMID 29628849
- [Background] Pai B H P, Shariat AN, Bhatt HV. PECS block for an ICD implantation in the super obese patient. J Clin Anesth. 2019 Nov;57:110-111. doi: 10.1016/j.jclinane.2019.04.003. Epub 2019 Apr 6. No abstract available. PMID 30965271
- [Background] Blanco R. The 'pecs block': a novel technique for providing analgesia after breast surgery. Anaesthesia. 2011 Sep;66(9):847-8. doi: 10.1111/j.1365-2044.2011.06838.x. No abstract available. PMID 21831090
- [Background] Hussain N, Brull R, McCartney CJL, Wong P, Kumar N, Essandoh M, Sawyer T, Sullivan T, Abdallah FW. Pectoralis-II Myofascial Block and Analgesia in Breast Cancer Surgery: A Systematic Review and Meta-analysis. Anesthesiology. 2019 Sep;131(3):630-648. doi: 10.1097/ALN.0000000000002822. PMID 31408448
- [Background] Bashandy GM, Abbas DN. Pectoral nerves I and II blocks in multimodal analgesia for breast cancer surgery: a randomized clinical trial. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):68-74. doi: 10.1097/AAP.0000000000000163. PMID 25376971
- [Background] Kulhari S, Bharti N, Bala I, Arora S, Singh G. Efficacy of pectoral nerve block versus thoracic paravertebral block for postoperative analgesia after radical mastectomy: a randomized controlled trial. Br J Anaesth. 2016 Sep;117(3):382-6. doi: 10.1093/bja/aew223. PMID 27543533